CLINICAL TRIAL: NCT05268640
Title: Comparison of the Efficacy of Emergency Double-level and Single Cervical Cerclage in Cervical Insufficiency in the Second Trimester of Pregnancy - Multicenter Prospective Randomized Trial
Brief Title: Cervical Occlusion Double-level Stitch Application
Acronym: COSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre of Postgraduate Medical Education (Other)
Collaborators: Polish Mother Memorial Hospital Research Institute (Other); Medical University of Warsaw (Other); Medical University of Gdansk (Other); Institute of Mother and Child, Warsaw, Poland (Other); Nicolaus Copernicus University in Toruń, Collegium Medicum in Bydgoszcz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: nr 1/2022
Record Dates: First submitted 2022-01-19; First posted 2022-03-07 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Cervical Incompetence
Keywords: pregnancy; premature birth; cervix; pregnancy complication
MeSH Terms: conditions — Uterine Cervical Incompetence; Premature Birth; Pregnancy Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Double-level cerclage (Experimental): double-level cervical cerclage placement with one suture above the other approximately 1 cm higher. Suture will be placed analogous to McDonald technique
  Interventions: Procedure: Double-level cervical cerclage
- Single-level cerclage (Active Comparator): single-level cervical cerclage of McDonald technique
  Interventions: Procedure: Single-level cervical cerclage

INTERVENTIONS:
Procedure: Double-level cervical cerclage — two cervical sutures + regimen of antibiotics + indomethacin + progesterone
  Arms: Double-level cerclage
Procedure: Single-level cervical cerclage — single cervical suture + regimen of antibiotics + indomethacin + progesterone
  Arms: Single-level cerclage

SUMMARY:
Cervical insufficiency is defined as painless dilatation of the cervix during the second trimester of pregnancy. As a result of shortening and opening of the cervix, despite the lack of uterine contractions, the fetal membranes invade into the cervical canal and then into the vagina, which results in premature rupture of the membranes and miscarriage or preterm delivery. Cervical insufficiency occurs in approximately 1% of the women. The aim of the study is to evaluate the effectiveness of placing a double-level cervical cerclage in the treatment of advanced cervical insufficiency. The hypothesis assumes that the insertion of a double-level suture is associated with a reduction in the rate of deliveries < 34 weeks of gestation in comparison to single-level suture. The study will include women with fetal membranes visible through open external os of the cervix between 16+0 and 25+6 weeks. They will be randomized to two arms - McDonald's single cervical cerclage or two-level cerclage.

DETAILED DESCRIPTION:
This is an open-label, multicentre, prospective, randomised controlled trial (RCT). Women will be randomized to the single-level cerclage arm or the double-level cerclage. Each patient will have a vaginal swab for aerobic and anaerobic bacteria and fungi culture, as well as for mycoplasmas, chlamydia and ureaplasma performed. Each patient will be treated with progesterone (vaginally 2 x 100 mg per day) and empirical antibiotic therapy (ceftriaxone 2.0 g iv + clarithromycin 2 x 500 mg po + metronidazole 3 x 500 mg iv for 7 days). If specific pathogens will be detected, the antibiotic therapy will be modified according to the antibiogram. If the diagnosis of cervical insufficiency will be made >23 weeks of gestation a single course of corticosteroid therapy will be administered (betamethasone 2 x 12 mg im) if the rsik of delivery within 7 days will be assessed as high. Indomethacin will also be administered for 48 hours (starting the day of cerclage administration, indomethacin 2 x 75 mg po for 48 hours). In the single-level cerclage arm McDonald suture will be administered. In the double-level cerclage arm two separate sutures analogous to McDonald technique will be placed, one approximately 1 cm higher above the other. Patients will be followed up until miscarriage or delivery and will receive standard perinatal care. Gestational age at delivery, the occurrence of cerclage complications and neonatal outcomes will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy,
* gestational age 16+0 to 25+6 weeks,
* live fetus,
* cervical incompetence with fetal membranes visible through external os before 24+0 weeks of gestation,
* informed written consent.

Exclusion Criteria - any of the following occuring before the administration of the cerclage:

* preterm premature rupture of membranes,
* vaginal bleeding,
* active regular uterine contractions,
* fetal demise,
* fever,
* intrauterine infection (diagnosed in case of maternal body temperature ≥ 38°C with no alternative cause identified and at least 2 symptoms among the following appear: fetal tachycardia > 160 bpm for 10 minutes or longer, uterine pain, purulent vaginal discharge, white blood cell count > 15 G/L in the absence of corticosteroid treatment or increased plasma C-reactive protein > 10 mg/L),
* known genetic defects of the fetus,
* known lethal fetal malformations,
* congenital uterine defects,
* multiple pregnancy.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female - pregnant women
Enrollment: 81 (Actual)
Dates: Start 2022-03-11 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
deliveries below 34+0 weeks of gestation | observation after intervention for 26 weeks of until birth
  number and rate of deliveries below 34+0 weeks of gestation

SECONDARY OUTCOMES:
gestational age at delivery | observation after intervention for 26 weeks of until birth
  duration of pregnancy untill delivery in weeks and days
time from cerclage administration to delivery | observation after intervention for 26 weeks of until birth
  time from cerclage administration to delivery in days
fetal demise | observation after intervention for 26 weeks of until birth
  number and rate of pregnancies complicated by fetal demise
neonatal outcomes | observation after intervention for 26 weeks of until birth
  number and rate of: congenital infections, respiratory morbidity, hospitalizations in the Neonatal Intensive Care Unit, early neurodevelopmental morbidity, gastrointestinal morbidity, retinopathy of prematurity, newborn's death before the discharge home
birth weight | observation after intervention for 26 weeks of until birth
  neonatal weight at delivery in grams
5th minute Apgar score | observation after intervention for 26 weeks of until birth
  neonatal general condition at 5th minute after delivery according to the Apgar Scale
maternal outcomes | observation after intervention for 26 weeks of until birth
  maternal mortality, miscarriage, intrauterine infection, prelabour rupture of membranes, o cervical laceration

OTHER OUTCOMES:
cerclage procedure complications occurring within 48 hours after cerclage placement | observation after intervention for 48 hours
  excessive vaginal bleeding, intrauterine infection, prelabour rupture of membranes

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna Kosinska Kaczynska, Prof., Principal Investigator — Center of Postgraduate Medical Education; Anna Kajdy, MD PhD, Principal Investigator — Center of Postgraduate Medical Education; Mariusz Grzesiak, Prof., Principal Investigator — Polish Mother's Memorial Hospital - Research Institute
Locations (7):
- Poland (7):
  - Department of Obstetrics, Women's Diseases and Oncological Gynecology, Nicolaus Copernicus University, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - 1st Department of Obstetrics and Gynecology, Center of Postagraduate Medical Education, Warsaw, Masovian Voivodeship
  - Department of Obstetrics, Perinatology and Neonatology, Center of Postagraduate Medical Education, Warsaw, Masovian Voivodeship
  - 1st Department of Obstetrics and Gynecology, Medical University of Warsaw, Warsaw, Masovian Voivodeship
  - Department of Obstetrics and Gynecology, Oncological Gynecology and Gynecological Endocrinology, Medical University of Gdansk, Gdansk, Pomeranian Voivodeship
  - Institute of Mother and Child, Warsaw
  - Polish Mother's Memorial Hospital - Research Institute, Lodz, Łódź Voivodeship

IPD SHARING:
Plan to Share IPD: Yes
IPD share with other researchers will include all IPD that underlie results in a publication
Supporting Information: Study Protocol, CSR
Time Frame: Data will become available after completing of recruitment and will be available for 12 months
Access Criteria: Data will be available od request sent to the principal researchers. All requests for information will be reviewed by the Study Officials.

REFERENCES:
- [Result] Daskalakis G, Papantoniou N, Mesogitis S, Antsaklis A. Management of cervical insufficiency and bulging fetal membranes. Obstet Gynecol. 2006 Feb;107(2 Pt 1):221-6. doi: 10.1097/01.AOG.0000187896.04535.e6. PMID 16449104
- [Result] Stupin JH, David M, Siedentopf JP, Dudenhausen JW. Emergency cerclage versus bed rest for amniotic sac prolapse before 27 gestational weeks. A retrospective, comparative study of 161 women. Eur J Obstet Gynecol Reprod Biol. 2008 Jul;139(1):32-7. doi: 10.1016/j.ejogrb.2007.11.009. Epub 2008 Feb 20. PMID 18243484
- [Result] Althuisius SM, Dekker GA, Hummel P, van Geijn HP; Cervical incompetence prevention randomized cerclage trial. Cervical incompetence prevention randomized cerclage trial: emergency cerclage with bed rest versus bed rest alone. Am J Obstet Gynecol. 2003 Oct;189(4):907-10. doi: 10.1067/s0002-9378(03)00718-x. PMID 14586323
- [Result] Oh KJ, Romero R, Park JY, Lee J, Conde-Agudelo A, Hong JS, Yoon BH. Evidence that antibiotic administration is effective in the treatment of a subset of patients with intra-amniotic infection/inflammation presenting with cervical insufficiency. Am J Obstet Gynecol. 2019 Aug;221(2):140.e1-140.e18. doi: 10.1016/j.ajog.2019.03.017. Epub 2019 Mar 28. PMID 30928565
- [Result] Miller ES, Grobman WA, Fonseca L, Robinson BK. Indomethacin and antibiotics in examination-indicated cerclage: a randomized controlled trial. Obstet Gynecol. 2014 Jun;123(6):1311-1316. doi: 10.1097/AOG.0000000000000228. PMID 24807330
- [Result] Wood SL, Owen J. Cerclage: Shirodkar, McDonald, and Modifications. Clin Obstet Gynecol. 2016 Jun;59(2):302-10. doi: 10.1097/GRF.0000000000000190. PMID 26974218
- [Result] Park JM, Tuuli MG, Wong M, Carbone JF, Ismail M, Macones GA, Odibo AO. Cervical cerclage: one stitch or two? Am J Perinatol. 2012 Jun;29(6):477-81. doi: 10.1055/s-0032-1304831. Epub 2012 Mar 7. PMID 22399222
- [Result] Giraldo-Isaza MA, Fried GP, Hegarty SE, Suescum-Diaz MA, Cohen AW, Berghella V. Comparison of 2 stitches vs 1 stitch for transvaginal cervical cerclage for preterm birth prevention. Am J Obstet Gynecol. 2013 Mar;208(3):209.e1-9. doi: 10.1016/j.ajog.2012.11.039. Epub 2012 Nov 28. PMID 23201330
- [Result] Woensdregt K, Norwitz ER, Cackovic M, Paidas MJ, Illuzzi JL. Effect of 2 stitches vs 1 stitch on the prevention of preterm birth in women with singleton pregnancies who undergo cervical cerclage. Am J Obstet Gynecol. 2008 Apr;198(4):396.e1-7. doi: 10.1016/j.ajog.2007.10.782. Epub 2008 Feb 21. PMID 18177834
- [Derived] Kosinska Kaczynska K, Rebizant B, Bednarek K, Dabrowski FA, Kajdy A, Muzyka-Placzynska K, Filipecka-Tyczka D, Uzar P, Kwiatkowski S, Torbe A, Grzesiak M, Kaczmarek P, Zyla M, Brawura-Biskupski-Samaha R. Emergency cerclage using double-level versus single-level suture in the management of cervical insufficiency (Cervical Occlusion double-level Stitch Application, COSA): study protocol for a multicentre, non-blinded, randomised controlled trial. BMJ Open. 2023 Jun 7;13(6):e071564. doi: 10.1136/bmjopen-2023-071564. PMID 37286317

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-01): https://cdn.clinicaltrials.gov/large-docs/40/NCT05268640/Prot_SAP_002.pdf
  • Informed Consent Form (2022-02-28): https://cdn.clinicaltrials.gov/large-docs/40/NCT05268640/ICF_003.pdf